CLINICAL TRIAL: NCT05266079
Title: Comparison Study of the Effectiveness Between Syndrome Differentiation Treatments and Fixed Formula Treatment for Perimenopausal Syndrome With Chinese Herbal Medicine
Brief Title: Comparison Study for Perimenopausal Syndrome With Chinese Herbal Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSPSCHM
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Menopausal Syndrome
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Syndrome differentiation treatment(GMBHDHT, TWBXD,SG,LWDHP and EZP, YGP and LZP) (Experimental): Syndrome differentiation treatment group of participants will be given medication by syndrome differentiating from qualified TCM Practitioners. TCM Practitioners will base on the syndrome of the participants to evaluate and modify the prescription after each assessment.
  1. Liver and Kidney Yin Deficiency syndrome use Gan Mai Bai He Di Hung Tang(GMBHDHT);
  2. Non Interaction Between Heart and Kidney syndrome use Tian Wang Bu Xin Dan(TWBXD);
  3. Liver Stagnation and Qi Stagnation syndrome use Shugan Granules(SG);
  4. Kidney Yin Deficiency syndrome use Liu Wei Di Huang Pill and Er Zhi Pill(LWDHP and EZP) ;
  5. Spleen and Kidney Yang Deficiency syndrome use You Gui pill and Li Zhong pill addition and subtraction(YGP and LZP).
  Each dose will be prepackaged in two identical foil sachets. Participants will be instructed to drink one sachet of granules dissolved in 200 mL of warm water twice daily.
  Interventions: Drug: Intervention Group
- Fixed formula treatment (Experimental): Fixed formula treatment Group will be given the standard formula Er-Xian decoction consisting of six herbs. The dosages of each herb were standardized according to the latest Chinese Medicine Recipe Dictionary (1997). The standard formula Er-Xian decoction are in the form of water-soluble granules. Each dose contains 11.8g and prepackaged in two identical foil sachets. Participants were instructed to drink one sachet of granules dissolved in 200 mL of warm water twice daily.
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Intervention Group — Gan Mai Bai He Di Hung Tang, Tian Wang Bu Xin Dan,Shugan Granules,Liu Wei Di Huang Pill and Er Zhi Pill , You Gui pill and Li Zhong pill addition and subtraction
  Other Names: Chinese herbal medicine
  Arms: Syndrome differentiation treatment(GMBHDHT, TWBXD,SG,LWDHP and EZP, YGP and LZP)
Drug: Control Group — Er-Xian decoction
  Other Names: Chinese herbal medicine
  Arms: Fixed formula treatment

SUMMARY:
Background: Perimenopausal syndrome (PMS) refers to a series of symptoms caused by the dynamic fluctuations of sex hormones during menopause. Menopausal symptoms including hot flushes, vaginal dryness and mood swings are experienced by about 80% of Chinese women aged 45 to 60. In the past year, 235 patients visited CMCTR(ND), a TCM center set up by HA and operated by HKFTU Workers' Medical Clinics since 2008, suffered from PMS.

According to literature review, high proportion of clinical trials regarding perimenopausal women used fixed formula treatment. However, different constitutional types were found in perimenopausal women and different fixed formulae were used in different research. Apart from kidney yin deficiency, perimenopausal women were also found in liver-kidney yin deficiency, kidney yang deficiency, kidney yin and yang deficiency, disharmony between heart and kidney, liver qi stagnation, etc. It is difficult to draw a conclusion that any single fixed formula could have the best efficacy on PMS. Therefore, it is worth studying to see whether syndrome differentiation would be a better choice for PMS treatment.

Objective: The study aims to evaluate whether syndrome differentiated treatment is better than fixed formula (Er-Xian decoction) treatment for perimenopausal women.

Design: This is a pilot single-blinded, randomized controlled trial.

Participants: Chinese women aged 45-55 year with menstruation abnormalities (menstrual irregularity in past 12 months; or menstrual period off at least twice in past 12 months; or amenorrhea of 2 to 12 months); also suffering any following perimenopausal symptoms: vasomotor symptoms (hot flushes, sweats), psychological symptoms (insomnia, migraine, irritability), or genitourinary symptoms (vaginal dryness, dyspareunia)

Interventions: A randomized controlled trial will be conducted to assess the efficacy of syndrome differentiated treatment versus a fixed formula (Er-Xian decoction) in treating PMS. 100 participants will be randomly divided into 2 groups. Intervention group of participants will be given medication by syndrome differentiating from qualified TCM Practitioners while the control group of participants will be given a fixed formula.

Outcome measures: Primary assessments outcome measure is the Kupperman Index, and the secondary outcome measure is MENQOL questionnaire.

DETAILED DESCRIPTION:
Perimenopausal syndrome is also known as menopausal syndrome. Menopause Syndrome refers to women due to ovarian dysfunction or loss of estrogen causing a variety of systemic dysfunctions in the body, including the autonomic nervous system, dysfunction and metabolic disorders-based symptoms such as hot flushes and sweating, sleep disorders, depression, multiple joint pains, headache, dizziness, fatigue, etc. These symptoms seriously affect menopausal women . Modern medical treatment of perimenopausal syndrome mainly focus on Hormonal Therapy (HT). Studies have shown that the clinical effect of hormonal therapy would quickly relieve the symptoms of perimenopausal syndrome, including urogenital atrophy and prevention of osteoporosis .

However there were some scholars believed that although short-term use of hormone supplement therapy could relieve the symptoms of perimenopausal women, the role of estrogen treatment in postmenopausal women still needed to be further explored . The reason was that hormonal replacement therapy can cause more adverse reactions and potential risks such as increased cardiovascular disease, cerebral infarction, breast-related diseases, risk of embolism in veins and lungs and other diseases .

In the previous study, the investigators found that the Chinese herbal formula Er-Xian decoction was superior to placebo in reducing the frequency and severity of hot flushes and in relieving menopausal symptoms in Hong Kong perimenopausal women. It was well tolerated, with no serious adverse events noted during the study period. The study proved the effectiveness of traditional Chinese medicine in the treatment of menopausal symptoms. The investigators designed this experiment in order to further understand the effectiveness between syndrome differentiation treatment and fixed prescription.

Syndrome differentiation and treatment is the process of recognizing and resolving diseases, the embodiment of the combination of theory and practice, the specific clinical application of principles and methods, and the basic principles guiding the clinical work of traditional Chinese medicine. Dialectics is the process of authentication. Syndrome is a summary of the pathological reflections of the body through four diagnostic methods (inspection, listening and smelling, inquiries, and palpation ). It would help to establish disease stages, including the location of disease, cause, nature, and relationship between healthy qi and pathogenic qi. Therefore, the syndrome would reveal the essence of the disease, and therefore enhance the disease management. Corresponding treatment method is determined based on the result of syndrome differentiation. Syndrome differentiation and treatment are two inseparable parts in the process of diagnosis and treatment of diseases.

There is no record of the term of the perimenopausal syndrome in the ancient Chinese medicine books. The investigators can find some similar symptoms recorded in "Lily Disease" , "Hysteria", and "Insomnia"or "Depression" and other diseases in ancient books. Modern Chinese medicine gynecology calls it "Premenopausal". Traditional Chinese medicine believes that in perimenopausal women, the kidney qi is gradually declining. Dysfunction of qi and blood is mainly caused by kidney deficiency. Among them, the syndrome of kidney yin deficiency is the most common. According to the literature, the syndrome types are divided as follows:

1. Liver and Kidney Yin Deficiency Syndrome: Before and after menstruation, the essence and blood are weak, or the body is in yin deficiency, yin does not guard the yang, yang is disturbed. Clinical symptoms include sweating, hot flushes, insomnia, forgetfulness, backache and weak legs, dry genitals, menstrual disorders, red tongue with less coating, pulse is rapid and thready. Suggested Formula: Gan Mai Bai He Di Hung Tang
2. Non Interaction Between Heart and Kidney:The woman's yin and yang are imbalanced, the yin essence is deficient, and the kidney yin deficiency and water does not nourish the wood, causing the liver fire to become prosperous. Common clinical symptoms include hot flush, sweating, palpitation, irritability, bitter mouth, dry mouth, red tongue with thin yellow coating, pulse is thready and rapid. Suggested formula: Tian Wang Bu Xin Dan
3. Liver stagnation and qi stagnation syndrome: Chest tightness, hypotension, chest pain, mental depression, nervousness, abdominal pain, flushing, nervousness, petechial, chord pulse. Suggested formula: Shugan Granules (Danzhi Xiaoyao San without Ginger add Xiangfu)
4. Kidney Yin Deficiency Syndrome: Fever, sweating, upset, Insomnia, dry mouth, ant feeling on the skin, early menstruation. Suggested formula: Liu Wei Di Huang Pill and Er Zhi Pill
5. Spleen and Kidney Yang Deficiency Syndrome:Fatigue, delayed menstruation, swelling, fear of cold, frequent urination, pale tongue, white fur, deep and thread pulse. Suggested formula: You Gui pill and Li Zhong pill addition and subtraction

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged 45-55 years
2. Menstruation abnormalities (menstrual irregularity in past 12 months; or menstrual period off at least twice in past 12 months; or amenorrhea of 2 to 12 months)
3. Suffering any of the following perimenopausal symptoms: vasomotor symptoms (hot flushes, sweats), psychological symptoms (insomnia, migraine, irritability), or genitourinary symptoms (vaginal dryness, dyspareunia)
4. Did not use hormonal therapy at least 3 months before entry into the study
5. Willing to give a written informed consent form to participate in the clinical study

Exclusion Criteria:

1. Bilateral ovarian resection or pelvic radiotherapy for ovarian cysts and uterine fibroids with a diameter greater than 4 cm
2. Unexplained irregular vaginal bleeding
3. Suffer from diabetic neuropathy or malignant tumor
4. Have used sex hormones in the past 3 months, such as estrogen, progesterone, soy isoflavones etc.
5. Patients who have participated in or are participating in other clinical trials in the past 3 months
6. Serious primary diseases such as cardiovascular, cerebrovascular, liver, kidney and hematopoietic system
7. Take sedatives or anti-anxiety drugs regularly
8. Smoking or alcohol habits
9. Patients with mental illness
10. Cannot cooperate with the treatment

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Kupperman Index | 8 weeks
  The evaluation is based on the clinical research experience of Kupperman HS in 1950s, which is composed of patient self-report and physician rating. The questionnaire includes 11 climacteric symptoms. The degree of symptoms was divide into four grades ranged from 0 to III: 0 for asymptomatic, I for occasional symptoms, II for frequent symptoms, and III for serious impact of life. These ratings were then summed across the 11 items and the score was categorized as follows: none 0-5, mild 5-10, moderate 10-15, severe 15+.

SECONDARY OUTCOMES:
Menopause Specific Quality of Life | 0,2,4,6,8,10,16 week
  Menopause Specific Quality of Life (MENQOL) was developed by Canadian scholars in 1996 as a tool to assess the quality of life of climacteric women. MENQOL is a self-management questionnaire. From the initial 106 items to 29 items, Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor, psychosocial, physical, and sexual. Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a zero (not bothersome) to six (extremely bothersome) scale. Means are computed for each subscale by dividing the sum of the domain's items by the number of items within that domain. For each item, participants are asked whether they have experienced each symptom in the past month and scored accordingly. The lower the score presents the higher the quality of life and the higher the score means the worse the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- HKFTU Workers' Medical Clinics - Hong Kong Baptist University Chinese Medicine Clinic cum Training and Research Centre (North District), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No